CLINICAL TRIAL: NCT02908698
Title: A Double-blind, Placebo-controlled Study to Evaluate the Effects of Oral Steroids on Skin of Patients With Moderate to Severe Atopic Dermatitis Patients
Brief Title: Effect of Oral Steroids on Skin Outcomes in Atopic Dermatitis
Acronym: OSAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary outcome was met in the 16 patients that completed the study per protocol
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Dr. Gail Gauvreau, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: McMaster-OSAD
Record Dates: First submitted 2016-09-08; First posted 2016-09-21 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone Treatment (Experimental): Prednisone will be administered orally for 15 days at the following doses:
  0.75 mg/kg of body weight for 5 days 0.5 mg/kg of body weight for 5 days 0.25 mg/kg of body weight for 5 days
  Interventions: Drug: Prednisone
- Placebo Control (Placebo Comparator): Placebo will be administered orally for 15 days in a capsule identical to the experimental treatment.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Prednisone — Total treatment duration: 15 days
  Doses are as follows:
  5 days daily treatment with 0.75 mg/kg of body weight 5 days daily treatment with 0.5 mg/kg of body weight 5 days daily treatment with 0.25 mg/kg of body weight
  Arms: Prednisone Treatment
Drug: Placebo Control — Total treatment duration: 15 days. Doses will appear identical to prednisone arm.
  Arms: Placebo Control

SUMMARY:
Atopic Dermatitis (AD), also known as eczema, is a common skin disease characterized by itchy lesions. The prevalence of AD has increased over the past few decades, with 15-30% of children and 2-10% of adults being affected. The lesions of atopic dermatitis patients are very inflamed, with an increased number of inflammatory cells in the skin. The first line treatment for AD is steroids, which reduce inflammation in the skin. There are several ways to measure if the treatment is effective, including clinical and cellular. We are proposing that a controlled skin allergen challenge will be an effective way to measure the effect of steroid at a cellular level through the measurement of inflammatory cells in the late cutaneous response. This will be examined using a placebo-controlled trial.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, parallel-group clinical trial to evaluate if steroid can block the late cutaneous response after intradermal allergen challenge. Individuals with moderate to severe atopic dermatitis that are develop late cutaneous response to intradermal allergen challenge will be eligible for enrollment. The study is divided into 2 parts.

Part 1: Screening

Subjects who meet all entry criteria will be screened with a medical history and physical examination. If they continue to meet entry criteria, their atopic status will be documented by skin testing against common airborne allergens (including cat, dust mite, grass, pollen) and an intradermal allergen challenge will be performed with a select allergen extract. Only subjects with a documented late cutaneous response to intradermal allergen challenge will be eligible for entry into Part 2 of the study.

Part 2: Dosing and Follow-up

Subjects will be randomly assigned 1:1 to receive either prednisone or placebo treatment. Prednisone treatment will be 5 days of 0.75 mg/kg, 5 days of 0.5 mg/kg and 5 days of 0.25 mg/kg. Before dosing and on Day 9 of dosing an intradermal allergen challenge will be performed and a skin biopsy of the late cutaneous response will be evaluated 24 hours after each intradermal allergen challenge. A sample of blood and skin from a lesion will be obtained before and on Day 9 of treatment. Patients will return for a follow up visit on Day 16 for safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18 through 65 years of age.
* Females must not be pregnant
* General good health
* Moderate to severe atopic dermatitis
* Able to understand and give written informed consent and sign a written informed consent form approved by the HIREB (Hamilton Integrated Research Ethics Board)
* Positive skin-prick test to common allergens (including cat, dust mite, grass, pollen)
* Positive late cutaneous response to intradermal allergen challenge

Exclusion Criteria:

* Treatment with an investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the baseline visit
* Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment:
* Immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, Interferon-γ (IFN-γ), Janus kinase inhibitors, azathioprine, methotrexate, etc.)
* Phototherapy for AD
* Treatment with biologics as follows:
* Any cell-depleting agents including but not limited to rituximab: within 6 months before the baseline visit, or until lymphocyte count returns to normal, whichever is longer
* Other biologics: within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever is longer
* Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (patients may continue using stable doses of such moisturizers if initiated before the screening visit)
* Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the baseline visit
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. Note: patients may be rescreened after infection resolves
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment
* History of human immunodeficiency virus (HIV) infection
* History of hepatitis B or hepatitis C infection
* Presence of skin comorbidities that may interfere with study assessments
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study
* Any other medical or psychological condition that may make patient's participation unreliable, or may interfere with study assessments.
* Planned or anticipated major surgical procedure during the patient's participation in this study
* Patient is a member of the investigational team or his/her immediate family
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Late Cutaneous Response (LCR) | Measured 24 hours after intradermal allergen challenge on day 2 and day 9 of study.
  Measured by size of the wheal.

SECONDARY OUTCOMES:
Comparison of eosinophils and basophils in the LCR between drug and placebo using histopathology. | Biopsy of LCR taken 24 hours after intradermal allergen challenge on day 2 and day 9 of study.
  The eosinophils and basophils will be measured by histopathology on the LCR biopsy.
Comparison of eosinophils and basophils in the LCR between drug and placebo using flow cytometry. | Biopsy of LCR taken 24 hours after intradermal allergen challenge on day 2 and day 9 of study.
  The eosinophils and basophils will be measured by flow cytometry on the LCR biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We plan to tabulate and include IPD in publication in medical journal.